CLINICAL TRIAL: NCT00132249
Title: A 40+ Year Post-Injury Follow-Up Study of Vietnam Veterans Who Sustained Traumatic Brain Injury While in Combat.
Brief Title: Vietnam Head Injury Study - Phase III
Status: Completed | Type: Observational
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); George Mason University (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); National Institutes of Health Clinical Center (CC) (NIH); University of York (Other); National Institute of Mental Health (NIMH) (NIH); University of Hertfordshire (Other); Georgetown University (Other); Cardiff University (Other)
Responsible Party: Sponsor
Other Study IDs: DAMD17-01-1-0675
Record Dates: First submitted 2005-08-17; First posted 2005-08-19 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Traumatic Brain Injury; Penetrating Head Injury; Closed Head Trauma
Keywords: Traumatic Brain Injury; Penetrating head wound; Closed head trauma; Vietnam Veteran
MeSH Terms: conditions — Brain Injuries, Traumatic; Head Injuries, Penetrating; Head Injuries, Closed

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Head Injured: The Vietnam Head Injured Subjects
- Head Uninjured: Uninjured Vietnam Veteran Control Subjects

SUMMARY:
The Vietnam Head Injury Study (VHIS)-Phase III is a prospective, long-term follow-up study of head-injured Vietnam veterans. The purpose of this research study is to determine the long-term consequences, if any, of head injury.

DETAILED DESCRIPTION:
The VHIS - Phase III evaluation to be conducted approximately 30 years post-injury will be devoted to examining, cutting-edge cognitive neuroscience issues and will utilize state of the art technologies to address basic research questions in the following areas: (1) Functions of the human prefrontal cortex; (2) Cognitive neuroplasticity in the aging brain; (3) Memory; (4) Long-term behavioral and psychosocial outcome; and (5) Neurological studies, including an evaluation of post-traumatic epilepsy and repeat clinical measures from Phase - II. This testing will be complemented with structural neuroimaging, electroencephalogram (EEG) and molecular genetics. The goals of the VHIS - Phase III include providing clinicians and scientists new insights into the long term recovery of function following brain injury, the role of the prefrontal cortex in executive functions, better predictors of long term outcome (including cognitive, neurological, and genetic factors), and the effects of head injury incurred in youth on aging and the development of dementia.

ELIGIBILITY:
The researchers are seeking healthy CONTROL participants.

Inclusion Criteria:

* Vietnam Veteran
* Served in active combat between 1966 - 1971
* Male

Exclusion Criteria:

* Any medical condition that would make participation detrimental to the control (i.e.: severe clinical depression, acute heart dysfunction, etc...)
* A history of severe head injury, stroke, loss of consciousness, or other significant neurological, psychiatric or medical condition that would render the subject unsuitable for the VHIS testing battery.

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 199 head-injured subjects attended PH3. 55 control subjects attended PH3.
Sampling Method: Probability Sample
Enrollment: 254 (Actual)
Dates: Start 2004-04; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
the assessment of a large number of the genetic markers and the relation to various out come measures. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Grafman, PhD, Principal Investigator — Cognitive Neuroscience Section, NINDS, NIH; Andres Salazar, MD, Principal Investigator — NINDS, NIH
Locations (1):
- National Naval Medical Center, Bethesda, Maryland, United States